CLINICAL TRIAL: NCT02088697
Title: A Bioequivalence Study of ASC-01 Placebo (Aripiprazole 0 mg/Sertraline 100 mg) and Sertraline Tablet in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 031-13-003
Record Dates: First submitted 2014-03-12; First posted 2014-03-17 (Estimated); Results first posted 2021-06-03 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Healthy Volunteers

ARMS (2):
- ASC-01 placebo (Experimental): A single oral dose of ASC-01 Placebo (sertraline 100 mg)
  Interventions: Drug: Placebo
- Sertraline tablet (Active Comparator): A single oral dose of sertraline tablets (sertraline 100 mg)
  Interventions: Drug: ASC-01

INTERVENTIONS:
Drug: Placebo
  Arms: ASC-01 placebo
Drug: ASC-01
  Arms: Sertraline tablet

SUMMARY:
The purpose of this study is to investigate the bioequivalence of ASC-01 Placebo and sertraline Tablet in Japanese healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers aged 20 to 40 years.
* Have a body mass index (BMI) between 18.5 and 25.0 kg/m2 and a weight of at least 50 kg.

Exclusion Criteria:

* History of any clinically important disease or disorder which, in the opinion of the Investigator, may either put the volunteer at risk because of participation in the study.
* History or presence of gastrointestinal, hepatic, or renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Any clinically significant abnormalities in the physical examination, clinical laboratory values, 12-lead ECG, or vital signs, as judged by the Investigator.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2013-12; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Osaka Pharmacology Clinical research Hospital, Osaka, Japan

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: ASC-01 Placebo First: Period I: A single oral dose of ASC-01 placebo (aripiprazole 0 mg/sertraline 100 mg) was administered after 10 or more hours of fasting.
  Period II: A single oral dose of sertraline tablets (sertraline 100 mg) was administered after 10 or more hours of fasting.
- Arm B: Sertraline First: Period I: A single oral dose of sertraline tablets (sertraline 100 mg) was administered after 10 or more hours of fasting.
  Period II: A single oral dose of ASC-01 placebo (sertraline 100 mg) was administered after 10 or more hours of fasting.
Period: Period I
Arm/Group | Arm A: ASC-01 Placebo First | Arm B: Sertraline First
Started | 25 | 25
Completed | 24 | 21
Not Completed | 1 | 4
Not completed — Physician Decision | 1 | 4
Period: Wash-out Period (at Least 10 Days)
Arm/Group | Arm A: ASC-01 Placebo First | Arm B: Sertraline First
Started | 24 | 21
Completed | 23 | 21
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Period II
Arm/Group | Arm A: ASC-01 Placebo First | Arm B: Sertraline First
Started | 23 | 21
Completed | 23 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: subjects who received the investigational medicinal product (IMP) at least once and from whom data on at least 1 safety endpoint were obtained after the start of IMP administration.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: ASC-01 Placebo First | Arm B: Sertraline First | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.2 (3.7) | 28.5 (4.3) | 26.8 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 25 | 25 | 50
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 25 | 25 | 50
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Peak Plasma Concentration (Cmax) of Sertraline
Time Frame: predose, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 144 and 168 hours postdose
Population: Bioequivalence Analysis Set comprised all subjects for whom the Cmax and AUCt were determined in both Period I and Period II.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- ASC-01 Placebo: A single oral dose of ASC-01 placebo (aripiprazole 0 mg/sertraline 100 mg) was administered after 10 or more hours of fasting.
- Sertraline: A single oral dose of sertraline tablets (sertraline 100 mg) was administered after 10 or more hours of fasting.
Arm/Group | ASC-01 Placebo | Sertraline
Number analyzed (Participants) | 44 | 44
ng/mL | 28.3 (8.31) | 28.8 (10.1)

2. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to the Last Observable Concentration at Time t (AUCt) for Sertraline
Time Frame: predose, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 144 and 168 hours postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | ASC-01 Placebo | Sertraline
Number analyzed (Participants) | 44 | 44
ng*h/mL | 835 (363) | 856 (421)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events occurring up to 8 days after dosing date were collected.
Description: A single dose of ASC-01 placebo or sertraline tablet was administered to 25 subjects each in Period I, and a single dose of ASC-01 placebo or sertraline tablet was administered to 21 and 23 subjects, respectively, in Period II. In this trial, safety data for each formulation were summarized based on subjects treated with the respective formulation, and safety was therefore evaluated in 46 subjects receiving ASC-01 placebo and 48 subjects receiving sertraline tablets.
Arm/Group | ASC-01 Placebo | Sertraline
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/48
Other Adverse Events (participants affected / at risk) | 9/46 | 19/48
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ASC-01 Placebo (N=46) | Sertraline (N=48)
Nausea (Gastrointestinal disorders) | 5 | 9
Diarrhoea (Gastrointestinal disorders) | 3 | 10
Vomiting (Gastrointestinal disorders) | 0 | 4
Blood bilirubin increased (Investigations) | 1 | 1
Blood sodium decreased (Investigations) | 1 | 2
Liver function test abnormal (Investigations) | 1 | 0
White blood cell count increased (Investigations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1
Eosinophil count increased (Investigations) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 1
Somnolence (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Ketonuria (Renal and urinary disorders) | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No